CLINICAL TRIAL: NCT06606769
Title: Fizyczne Aktywnosci Gwarantem Zdrowych Kosci
Brief Title: Physical Activity Guarantees Bone Density.
Acronym: BONES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RO_NdS_MNiSW2024; NdS-II/SP/0364/2023/01 (Other Grant/Funding Number: Polish Ministry of Science and Higher Education)
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Osteoporosis; Osteopenia
Keywords: physical activity; bone mineral density
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- exercise (Experimental): supervised exercise training; twice a week for 12 months
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — supervised exercise training; twice a week for 12 months

SUMMARY:
Bone tissue is crucial for overall health and quality of life, but it undergoes constant internal remodeling, leading to osteoporosis, a widespread bone disease. Regular physical activity can improve bone mineral density (BMD) and prevent osteoporosis. Studies have shown that premenopausal women with regular physical activity have greater BMD. Diagnosing bone resorption is essential, and dual-energy X-ray absorptiometry tests (DXA) and circulating microRNAs (miRNAs) may offer more prognostic potential than conventional markers. The gut microbiome may also regulate bone metabolism, with metabolites like trimethylamine N-oxide (TMAO) playing a role. A project aims to promote systematic physical activity to improve BMD and well-being, support societal mobilization, and conduct preventive examinations for osteoporosis risk. Implementing systematic prevention is important not only for health but also for reducing social and financial costs associated with osteoporosis and associated fractures.

DETAILED DESCRIPTION:
Bone tissue, in addition to providing the body with supportive functions and protecting organs from injury, is a metabolically active tissue that influences the proper functioning of other organs. Therefore, bones are essential for overall health and quality of life. Bones undergo constant internal remodeling. With prolonged resorption dominance, bone mass decreases, accompanied by a deterioration of microarchitecture leading to impaired bone strength. This pathological condition is called osteoporosis and is one of the most widespread bone diseases in the world.

In recent years, there has been increasing discussion about the beneficial impact of physical activity on human health. Broadly understood physical activity affects the skeletal system, which translates into the stimulation of processes related to bone formation in the body. It is very important that exercises are performed regularly. Among premenopausal women who regularly engage in physical activity, a greater bone mineral density (BMD) has been observed compared to a group of women who do not participate in any physical activity. Therefore, there is a need to promote physical activity and to tailor physical activities according to the needs arising from both the principles of osteoporosis prevention and the age or hormonal status of women.

It is important to note that bone tissue loss is painless and progresses asymptomatically, gradually weakening the bones. Therefore, it is very important to conduct studies that diagnose the progress of bone resorption. A milestone in the diagnosis of osteoporosis is undoubtedly the dual-energy X-ray absorptiometry test. (DXA). Circulating microRNAs (miRNAs) may potentially serve as an attractive alternative or addition to the diagnostic arsenal and offer greater prognostic potential than conventional markers. Furthermore, an increasing number of studies show that the gut microbiome may be a key factor regulating bone physiology. It has been shown that bone metabolism can be regulated by metabolites dependent on the gut microbiome. The metabolite in question is trimethylamine N-oxide. (TMAO). However, so far, there have been few studies addressing the impact of TMAO on bone metabolism, as well as the underlying molecular mechanisms, and the results obtained are not conclusive.

The project aims to promote systematic physical activity that improves not only BMD but also the well-being of every individual who exercises. By increasing the availability of activation programs, this project supports the mobilization of society. Furthermore, the preventive examinations conducted among individuals qualified for the project allow for the early detection of an increased risk of developing osteoporosis. Early diagnosis of the disease prevents serious consequences in the future and increases the chances of a complete cure. At the same time, the project will undertake pioneering research aimed at enhancing the quality and excellence of the scientific and research staff.

The implementation of systematic prevention for this condition is particularly important not only in the context of health but also due to the significant social and financial costs of treating the consequences of osteoporosis and its associated fractures.

ELIGIBILITY:
Inclusion Criteria:

women

Exclusion Criteria:

diagnosed osteoporosis

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
bone mineral density | before and after 12 months of intervention
  BMD using dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
blood markers | before and after 12 months of intervention
  C-terminal telopeptide of type 1 collagen aminoterminal propeptide of type I procollagen trimethylamine N-oxide microRNA complete blood count
physical fitness tests | before and after 12 months of intervention
  hand grip strength maximum vertical jump Chester step test

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Olek, professor, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No
we will consider sharing individual participant data in the future